CLINICAL TRIAL: NCT04385888
Title: Effects of Low-calorie Sweetened Beverage Restriction in Youth With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allison Sylvetsky (Meni) (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor-Investigator, Allison Sylvetsky (Meni), Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00012436
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-calorie sweetener restriction (Experimental): Participants will be instructed to avoid low-calorie sweetened beverages and other sources of low-calorie sweeteners, and to instead consume unsweetened alternatives, such as plain or sparkling water for 12 weeks.
  Interventions: Behavioral: Low-calorie sweetener restriction
- Usual consumption/control (No Intervention): Participants will continue low-calorie sweetener consumption, as usual.

INTERVENTIONS:
Behavioral: Low-calorie sweetener restriction — Participants will avoid low-calorie sweetened beverages and other sources of low-calorie sweeteners for 12 weeks and will instead consume unsweetened alternatives, such as still or sparkling water
  Arms: Low-calorie sweetener restriction

SUMMARY:
This study will investigate whether low-calorie sweeteners (LCS) are helpful or harmful for preventing diabetes complications among children with Type 1 Diabetes (T1D).

DETAILED DESCRIPTION:
Eligible participants will be scheduled for a baseline visit. During the week prior, they will be instructed to continue usual dietary habits and complete an online photo-assisted food record, with parental assistance. At the baseline visit, height and weight will be measured, a spot urine sample will be collected, and a blood draw will be performed. Participants will have their CGM data for the past two weeks downloaded. In a subset of participants, an abdominal MRI will also be performed.

Subjects will then be randomized to either: 1) low-calorie sweetener (LCS) restriction or 2) continuation of usual LCS intake (control). All participants (both groups) and their parent will undergo a brief, 20-minute orientation where the PI and study dietitian will provide an introduction to the study, instructions on completing food records, education on CGM. Those in the intervention group will be given sample replacement beverages and a brochure on avoiding LCS to take home which will include a list of specific foods and beverages containing LCS to avoid during the study. Participants in the control group will be counseled on healthy eating as those in the intervention group (in accordance with standard dietary guidance for T1D management), with the exception of information and resources for avoiding LCS.

In both groups, text messages will be sent to parents 3X/week with reminders that their child should avoid LCS or continue usual intake, per randomization. Adherence will be monitored through collection of spot-urine samples for measurement of sucralose and ace-K concentrations. daily text message beverage logs completed by the parent, and photo-assisted food records with parent assistance in Weeks 0, 1, 6, and 12. During Week 6, participants and their parent will attend a mid-intervention telemedicine booster visit, during which the PI and/or study RA will reinforce the intervention and remind participants to mail back a spot urine sample using materials provided by the study team at baseline. Participants will be reminded of the study instructions, including the importance of inserting the DEXCOM G6 sensor (provided by study team) at the beginning of Week 11.

At the end of Week 12, participants and their parent will return for follow-up. Participants will have their CGM data downloaded using DEXCOM Clarity™ software. Height and weight will be measured and a second blood draw performed. Those who had an MRI at the baseline visit (n=30) will undergo a second abdominal MRI. Those randomized to the intervention will be purposefully sampled and asked to complete a ~20 minute qualitative interview and ~5 minute satisfaction survey, together with their parent, about their study experience and the challenges of LCSB restriction.

ELIGIBILITY:
Inclusion Criteria:

1. Child 6-12 years old
2. Report consumption of ≥ 12 oz. beverages with sucralose (+/- ace-K) or aspartame+ace-K per day
3. Child has had a diagnosis of T1D for at least one year
4. Parent/guardian has reliable phone and internet access
5. Parent/guardian and child both speak English
6. Child is enrolled in the Diabetes Program at Children's National Hospital

Exclusion Criteria:

1. Child under 6 years of age
2. Child older than 12 years of age
3. Child consumes foods with low-calorie sweeteners more than 3 times per week
4. Child consumes condiments with low-calorie sweeteners more than 3 times per week
5. Child has poorly managed chronic disease other than T1D or is taking medications other than insulin

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sylvetsky AC, Moore HR, Kaidbey JH, Halberg SE, Cogen FR, DiPietro L, Elmi A, Goran MI, Streisand R. Rationale and design of DRINK-T1D: A randomized clinical trial of effects of low-calorie sweetener restriction in children with type 1 diabetes. Contemp Clin Trials. 2021 Jul;106:106431. doi: 10.1016/j.cct.2021.106431. Epub 2021 May 8. PMID 33974993

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reason that the number started does not equal the total enrollment is because there was a run-in period, prior to randomization, where 3 children (6 total participants including the child's parent) were lost to follow-up.
Groups:
- Low-calorie Sweetener Restriction: Children: Participants will be instructed to avoid low-calorie sweetened beverages and other sources of low-calorie sweeteners, and to instead consume unsweetened alternatives, such as plain or sparkling water for 12 weeks.
  Low-calorie sweetener restriction: Participants will avoid low-calorie sweetened beverages and other sources of low-calorie sweeteners for 12 weeks and will instead consume unsweetened alternatives, such as still or sparkling water
- Usual Consumption/Control: Children: Participants will continue low-calorie sweetener consumption, as usual.
- Low-calorie Sweetener Restriction: Parents: Participants will be instructed to have their child avoid low-calorie sweetened beverages and other sources of low-calorie sweeteners, and to instead consume unsweetened alternatives, such as plain or sparkling water for 12 weeks.
- Usual Consumption/Control: Parents: Participants'children will continue low-calorie sweetener consumption, as usual.
Period: Run-in Period
Arm/Group | Low-calorie Sweetener Restriction: Children | Usual Consumption/Control: Children | Low-calorie Sweetener Restriction: Parents | Usual Consumption/Control: Parents
Started | 16 | 15 | 16 | 15
Completed | 15 | 13 | 15 | 13
Not Completed | 1 | 2 | 1 | 2
Period: Randomized to Intervention or Control
Arm/Group | Low-calorie Sweetener Restriction: Children | Usual Consumption/Control: Children | Low-calorie Sweetener Restriction: Parents | Usual Consumption/Control: Parents
Started | 15 | 13 | 15 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were not collected for parents.
Groups:
- Usual Consumption/Control: Parents: Participants' children will continue low-calorie sweetener consumption, as usual.
- Total: Total of all reporting groups
Arm/Group | Low-calorie Sweetener Restriction: Children | Usual Consumption/Control: Children | Low-calorie Sweetener Restriction: Parents | Usual Consumption/Control: Parents | Total
Number analyzed (Participants) | 15 | 13 | 0 | 0 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (1.8) | 9.7 (2.3) |  |  | 9.7 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 |  |  | 14
  Male | 8 | 6 |  |  | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 |  |  | 2
  Not Hispanic or Latino | 14 | 12 |  |  | 26
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 0 | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 6 | 6 |  |  | 12
  White | 8 | 6 |  |  | 14
  More than one race | 1 | 1 |  |  | 2
  Unknown or Not Reported | 0 | 0 |  |  | 0
BMI percentile [Mean (Standard Deviation); unit: percentile] | 62.1 (29.0) | 73.9 (15.0) |  |  | 67.6 (23.9)
Time since type 1 diabetes diagnosis [Mean (Standard Deviation); unit: years] | 4.0 (2.9) | 4.4 (2.1) |  |  | 4.2 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Variability
Description: Change in Time in Range (TIR)
Time Frame: Baseline vs Weeks 11-12
Population: The outcome was measured only among children who completed the study.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Low-calorie Sweetener Restriction | Usual Consumption/Control | Low-calorie Sweetener Restriction: Parents | Usual Consumption/Control: Parents
Number analyzed (Participants) | 13 | 13 | 0 | 0
percent | 2.00 (2.59) | 3.91 (2.59) |  |

2. Secondary Outcome: Visceral Adiposity
Description: Change in visceral fat area will be assessed using DXA. Due to COVID-19, very few participants were able to have visceral fat measured pre and post intervention.
Time Frame: Baseline vs. Week 12
Population: Outcomes were assessed for children, not parents
Measure: Mean (Standard Error); unit: % body fat
Arm/Group | Low-calorie Sweetener Restriction | Usual Consumption/Control | Low-calorie Sweetener Restriction: Parents | Usual Consumption/Control: Parents
Number analyzed (Participants) | 3 | 5 | 0 | 0
% body fat | 0.1 (1.1) | 1.0 (0.8) |  |

3. Secondary Outcome: Change in Inflammatory Cytokines (TNF-alpha)
Description: We will collect a blood sample to measure TNF-alpha and calculate the change from baseline.
Time Frame: Baseline vs Week 12
Population: The outcome was measured among children, not parents.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low-calorie Sweetener Restriction | Usual Consumption/Control | Low-calorie Sweetener Restriction: Parents | Usual Consumption/Control: Parents
Number analyzed (Participants) | 13 | 13 | 0 | 0
pg/mL | 0.08 (0.07) | -0.23 (0.08) |  |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant during the 14 weeks they were enrolled in the study.
Groups:
- Low-calorie Sweetener Restriction: Parents: Participants were instructed to have their child avoid low-calorie sweetened beverages and other sources of low-calorie sweeteners, and to instead consume unsweetened alternatives, such as plain or sparkling water for 12 weeks.
Arm/Group | Low-calorie Sweetener Restriction: Children | Usual Consumption/Control: Children | Low-calorie Sweetener Restriction: Parents | Usual Consumption/Control: Parents
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/15 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT04385888/Prot_SAP_000.pdf